CLINICAL TRIAL: NCT05509023
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 2a Proof-of-Concept Study Evaluating the Safety and Efficacy of ADX-914 in Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: Evaluating Safety and Efficacy of ADX-914 in Patients With Moderate to Severe Atopic Dermatitis (SIGNAL-AD)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Q32 Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ADX-914-202
Record Dates: First submitted 2022-08-12; First posted 2022-08-19 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Eczema Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ADX-914 (Experimental)
  Interventions: Drug: ADX-914
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ADX-914 — Subcutaneous administration of ADX-914
  Arms: ADX-914
Drug: Placebo — Subcutaneous administration of Placebo
  Arms: Placebo

SUMMARY:
This is a phase IIa, randomized, double-blind, placebo-controlled, multi-center proof-of-concept (POC) study in subjects with moderate to severe Atopic Dermatitis.

DETAILED DESCRIPTION:
This is a two-part phase IIa, randomized, double-blind, placebo-controlled, multi-center proof-of-concept (POC) study in adult subjects with persistent moderate to severe Atopic Dermatitis (AD). ADX-914 or matching placebo for administered subcutaneously in the clinic setting every 2 weeks for 12 weeks, and follow-up for 12 weeks. ADX-914 or matching placebo will be in the clinic setting post-randomization. In Part A, up to 3 cohorts of subjects will be randomized 2:1 drug vs placebo. In Part B subjects will be randomized 1:1 to drug vs placebo at a doses selected in Part A.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, inclusive, at time of informed consent, with chronic AD (duration of disease ≥3 years) diagnosed by the Eichenfield revised criteria of Hanifin and Rajka.
2. Moderate to severe disease activity at baseline and screening defined as:

   1. BSA affected ≥10%
   2. EASI Score ≥12
   3. Investigators Global Score (IGA) ≥3
3. Who, in the opinion of the Investigator, have a history of inadequate response to at least one of the following:

   1. at least 4-week course of medium-potency topical steroids or other approved topical immunomodulators (calcineurin, PDE-4 and JAK inhibitors)
   2. systemic steroids or phototherapy
   3. oral chemical synthetic immunomodulators (MTX, mycophenolate mofetil, azathioprine, cyclosporine, systemic approved biologics [dupliumab, ustekinumab or tralokinumab]), or approved systemic targeted synthetic JAK inhibitors (upadacitinib, abrocitinib)

Exclusion Criteria:

1. Body weight ≤ 50.0 kg for men and ≤ 45.0 kg for women and > 120 kg at Screening
2. Rescue therapy, topical or systemic, need anticipated within 4 weeks of randomization
3. Recent (within 2 months of informed consent) or current clinically serious viral, bacterial, fungal, or parasitic infection or mycobacterial infection
4. A positive QuantiFERON®TB Gold test at Screening or history of tuberculosis (TB)
5. Have been exposed to a live vaccine within 12 weeks prior to planned randomization or are expected to receive a live vaccine during the study
6. Systemic, topical or device-based therapy of AD
7. Serious concomitant illness that could require the use of systemic corticosteroids or otherwise interfere with study participation or require active frequent monitoring
8. Other concomitant skin conditions that would interfere with evaluations of the effect of study medication on atopic dermatitis
9. Other active autoimmune diseases other than those above that would make it difficult to appropriately assess AD disease activity or pose a risk to the subject's participation in the trial
10. Pregnant or lactating women, or women planning to become pregnant or initiate breastfeeding.
11. History of sensitivity to any of the study treatments, or components thereof, or a history of drug or other allergy that, in the opinion of the Investigator, contraindicates their participation.
12. Has been in another investigational trial within 30 days or 5 half-lives of the investigational agent (whichever is greater) prior to the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Part A only: Safety parameters including incidence of serious adverse events and adverse events of special interest | 14 Weeks
Part A and B: Mean percentage change from baseline in Eczema Area and Severity Index (EASI) score at Week 14 for ADX-914 vs placebo | 14 Weeks
  Severity score is based on evaluation of severity of atopic dermatitis in 4 body regions (head and neck, trunk, upper limbs, and lower limbs). The minimum score is 0 (less severe) and maximum score is 72 (most severe).

SECONDARY OUTCOMES:
Mean percentage change from baseline in Eczema Area and Severity Index (EASI) score | 24 Weeks
  Severity score is based on evaluation of severity of atopic dermatitis in 4 body regions (head and neck, trunk, upper limbs, and lower limbs). The minimum score is 0 (least severe) and maximum score is 72 (most severe)
Mean percentage change from baseline in Scoring Atopic Dermatitis (SCORAD) score | 24 Weeks
  Score is based on evaluation of 6 body regions (Head and neck, upper limbs, lower limbs, anterior trunk, back, and genitals). The minimum score is 0% (least severe) and the maximum score is 100% (most severe)
Proportion of subjects achieving Eczema Area and Severity Index (EASI) reduction of 50%, 75% and 90% | 24 Weeks
  Severity score is based on evaluation of severity of atopic dermatitis in 4 body regions (head and neck, trunk, upper limbs, and lower limbs). The minimum score is 0 (least severe) and maximum score is 72 (most severe)
Proportion of subjects achieving Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) score of 0 or 1 with at least 2 grades of reduction from Baseline | 24 Weeks
  Score is based on Investigator's impresion of the severity of Atopic Dermatitis with 0 being the least severe and 4 being the most severe
Incidence of adverse events | 24 Weeks
  As evaluated by vital signs, physical examinations, laboratory evaluations, and 12-lead electrocardiograms

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Cahaba Dermatology Skin Health Center, Birmingham, Alabama
  - First OC Dermatology, Fountain Valley, California
  - California Allergy and Asthma Medical Group- Los Angeles, Los Angeles, California
  - Integrative Skin Science and Research, Sacramento, California
  - Dermatology Institute and Skin Care Center, Santa Monica, California
  - Torrance Clinical Research Institute Inc., Torrance, California
  - Integrated Research of Inland, Inc., Upland, California
  - RM Medical Research Inc., Homestead, Florida
  - Medical Research Center of Miami, Miami, Florida
  - Well Pharma Medical Research Corporation, Miami, Florida
  - GCP Research, St. Petersburg, Florida
  - Advanced Medical Research, PC, Sandy Springs, Georgia
  - Treasure Valley Medical Research, Boise, Idaho
  - Sneeze wheeze and Itch Associates LLC, Normal, Illinois
  - Southern Indiana Clinical Trials, New Albany, Indiana
  - Visage Clinical Research, Largo, Maryland
  - Revival Research Corporation- Clinedge, Troy, Michigan
  - Apex Clinical Research Center, Painesville, Ohio
  - Clinical Partners, LLC, Johnston, Rhode Island
  - North Texas Center for Clinical Research, Frisco, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - JBR Clinical Research, Salt Lake City, Utah
  - Dermatology of Seattle & Bellevue, Seattle, Washington
  - Dermatology Specialists of Spokane, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No